CLINICAL TRIAL: NCT02140606
Title: An Open Phase I Trial to Investigate the Maximum Tolerated Dose, Safety, Pharmacokinetics, and Efficacy of Intravenous Cafusertib Hydrochloride in Combination With Subcutaneous Low Dose Cytarabine in Chinese Patients With Acute Myeloid Leukaemia (AML)
Brief Title: Phase I Trial to Investigate Cafusertib Hydrochloride in Combination With Low Dose Cytarabine in Chinese Patients With Acute Myeloid Leukaemia (AML)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10159-I-01
Record Dates: First submitted 2014-05-12; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML; phase1; MTD; Cafusertib
MeSH Terms: conditions — Leukemia, Myeloid, Acute

ARMS (1):
- Cafusertib Hydrochloride + Cytarabine (Experimental): Cafusertib (d1 and 15 - one hour iv.) + LD ARA C 2x20 mg/d s.c. Patient to receive escalating dose of cafusertib hydrochloride.
  Interventions: Drug: Cafusertib Hydrochloride

INTERVENTIONS:
Drug: Cafusertib Hydrochloride — Drug: Cafusertib Hydrochloride (d1 and 15) Cafusertib (d1 and 15 - one hour iv.v) Drug: Cytarabine Cytarabine 2 x 20 mg/d s.c. d1-15.

SUMMARY:
To investigate safety, tolerability of cafusertib combination with low dose cytarabine (LD-Ara-C) in Chinese patients with relapsed/refractory AML that are not eligible for conventional or intensive treatment. The dose of cafusertib will be escalated to determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) of cafusertib in combination with LD-Ara-C in AML patients. At the same time, pharmacokinetic characteristics and preliminary efficacy of cafusertib will be observed in AML patients. To determine the recommended dosage regimen for phase II.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent consistent with Chinese Good Clinical Practice.
* Male or female patients of age >/= 18 years at the time of informed consent.
* Patients with relapsed/refractory AML ineligible for conventional or intensive treatment.
* Eastern Cooperative Oncology Group performance status score 0 - 2 at screening.
* Life expectancy of at least 3 months.
* Adequate hepatic, renal and metabolic function parameters: Serum total bilirubin ≤1.5 x upper limit of normal, aspartate transaminase (AST) , alanine transaminase (ALT) ≤2.5 x upper limit of normal; Creatinine clearance rate ≥60ml/min, Serum creatinine ≤1.0 x upper limit of normal; Relatively normal ECG(electrocardiogram), QTc<450 ms(male) ,QTc<470 ms(female); LVEF>50%.
* Patients who can comply with the trial and follow-up procedures.

Exclusion Criteria:

* Patients had received cafusertib hydrochloride or other PLK inhibitors.
* Patients with APL.
* Patients with central nervous system leukemia.
* Need to continue using cytokine therapy at screening.
* Patients participated in other clinical trials within 4 weeks prior to enrollment.
* Patient with severe infection.
* Patients with myocardial infarction had occurred within six months prior to enrollment.
* Severe heart disease, including NYHA class II cardiac dysfunction and above.
* Patients with HIV infection or acute and chronic viral hepatitis.
* Severe gastrointestinal disorders (bleeding, infection, obstruction or greater than grade 1 diarrhea).
* A previous history of neurological or psychiatric disorders, including epilepsy or dementia.
* Concomitant medications with CYP3A4 inhibitors, inducers or substrates; Women pregnant or breast feeding.
* Subject is thought unfit for this study by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
MTD of cafusertib in combination with LDAraC based on the incidence of dose limiting toxicities | 4 weeks

SECONDARY OUTCOMES:
Efficacy (complete remission, CR; complete remission with incomplete blood count recovery, Cri; Partial remission (PR)) | minimum 4 weeks, maximum n.a.
Incidence and intensity of adverse events graded according to CTCAE (version 4.0) | minimum 4 weeks, maximum n.a.
Incidence of dose limiting toxicity (DLT) | 4 weeks
Pharmacokinetics of cafusertib | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Blood Diseases, Chinese Academy of Medical Sciences, Tianjin, China